CLINICAL TRIAL: NCT00506441
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-center, Withdrawal Study Comparing MCI-196 v.s Placebo Following A 12-Week Dose Titration Period With MCI-196 in Stage V Subjects on Dialysis With Hyperphosphatemia
Brief Title: A Phase 3, Randomized, Double Blind, Placebo-Controlled, Multi-Center, Withdrawal Study of MCI-196 in CKD on Dialysis With Hyperphosphatemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCI-196-A05
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Results first posted 2014-07-25 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease; Dialysis; Hyperphosphatemia
Keywords: Chronic Kidney Disease; Dialysis; Hyperphosphatemia; Phosphate binder
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — cholebine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: MCI-196
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MCI-196 — 3g to 15g/day (3 times a day), Tablet, 12 weeks of flexible dose (Open-label) and 4 weeks of double blind
  Other Names: Colestilan(INN); Colestimide(JAN); CHOLEBINE®; BindRen®
  Arms: 1
Drug: Placebo — 3g to 15g/day (3 times a day), Tablet, 4 weeks of double blind
  Arms: 2

SUMMARY:
This is a phase III multi-centre study in three periods: the first period is a phosphate binder washout for 4 weeks, the second period is an open-label, flexible dose titration, the third period is a placebo-controlled withdrawal comparing MCI-196 with placebo for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, and is >=18 years old
* Stable hemodialysis or peritoneal dialysis
* Subjects has Stable phosphate control
* Subjects on Stabilized phosphorus diet
* Subjects undergoing regular dialysis treatment
* Female and of child-bearing potential have a negative serum pregnancy test.
* Male subjects must agree to use appropriate contraception.

Exclusion Criteria:

* Current clinically significant medical comorbidities, which may substantially compromise subject safety, or expose them to undue risk, or interfere significantly with study procedures and which, in the opinion of the Investigator, makes the subject unsuitable for inclusion in the study.
* serum albumin level < 3.0g/dL
* PTH level > 1000pg/mL
* Hemoglobin level < 8mg/dL
* A History of significant gastrointestinal motility problems
* Biliary obstruction or proven liver dysfunction
* A positive test for hepatitis B surface antigen, hepatitis C antibody or HIV 1 and 2 antibodies
* A clinically significant severe lactose intolerance or sensitivity
* A history of substance or alcohol abuse within the last year.
* Seizure disorders
* A history of drug or other allergy
* using cholestyramine, colestipol or colesevelam
* Schedule to receive a kidney transplant within the next 6 months
* Participation in a clinical study with any experimental medication in the last 30 days or an experimental biological product within the last 90 days prior to signing of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Principal Investigator — Information at Mitsubishi Pharma America
Locations (39):
- United States (38):
  - Glendale, Arizona
  - Tempe, Arizona
  - Hot Springs, Arkansas
  - Paragould, Arkansas
  - Pine Bluff, Arkansas
  - Fountain Valley, California
  - La Mesa, California
  - Long Beach, California
  - Lynwood, California
  - Orange, California
  - San Diego, California
  - Whittier, California
  - Brandon, Florida
  - Hudson, Florida
  - Lauderdale Lakes, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Decatur, Georgia
  - Macon, Georgia
  - Evanston, Illinois
  - Evergreen Park, Illinois
  - Fort Wayne, Indiana
  - Shreveport, Louisiana
  - Springfield, Massachusetts
  - Eatontown, New Jersey
  - Flushing, New York
  - Springfield Gardens, New York
  - Allentown, Pennsylvania
  - Lewistown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Orangeburg, South Carolina
  - Sumter, South Carolina
  - San Antonio, Texas
  - Alexandria, Virginia
  - Portsmouth, Virginia
  - Richmond, Virginia
  - West Allis, Wisconsin
- San Juan, Puerto Rico

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Hertel J, Locatelli F, Spasovski G, Dimkovic N, Wanner C. Randomized, Double-Blind, Placebo-Controlled, Withdrawal Study of Colestilan after Dose Titration in Chronic Kidney Disease Dialysis Patients with Hyperphosphatemia. Nephron. 2015;130(4):229-38. doi: 10.1159/000431289. Epub 2015 Jul 10. PMID 26184491

RESULTS

PARTICIPANT FLOW:
Groups:
- MCI-196: Open-label Period (Week 0 -12) ; 3, 6, 9, 12, or 15 g/ day as titrated
  Double-blind Period (Week 12 - 16) ; dose level at the end of dose titration in the Open-label period
- Placebo: Double-blind Period (Week 12 - 16) ; dose level at the end of dose titration in the Open-label period
Period: Period 1; Open-label Period
Arm/Group | MCI-196 | Placebo
Started | 245 | 0
Completed | 169 | 0
Not Completed | 76 | 0
Not completed — Adverse Event | 21 | 0
Not completed — Lack of Efficacy | 13 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 5 | 0
Not completed — Protocol Violation | 9 | 0
Not completed — Withdrawal by Subject | 13 | 0
Not completed — Other Reasons | 13 | 0
Period: Period 2; Double-blind Period
Arm/Group | MCI-196 | Placebo
Started | 85 | 84
Completed | 82 | 79
Not Completed | 3 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other Reason | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- MCI-196: Open-label Period (Week 0 - 12) ; 3, 6, 9, 12, or 15 g/ day as titrated
  Double-blind Period (Week 12 - 16) ; dose level at the end of dose titration in the Open-label period
Arm/Group | MCI-196
Number analyzed (Participants) | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 146

OUTCOME MEASURES:

1. Primary Outcome: The Change in Serum Phosphorus From Week 12 to Week 16
Description: The changes in serum phosphorus (mg/dL) from Week 12 to Week 16 (last observation post Week 12)
Time Frame: 4 weeks (Week 12 to Week 16)
Population: Intent-to-treat (ITT) 2 (The ITT2 population included all subjects who complete 12-weeks, receive a randomization number and receive at least one dose of study medication in the placebo-controlled withdrawal phase, either MCI-196 or placebo, and have at least one central phosphorus value after 12-weeks.)
Measure: Mean (Standard Deviation); unit: mg / dL
Groups:
- MCI-196 (Double-blind Period); Placebo (Double-blind Period): Double-blind Period (Week 12 - 16) ; dose level at the end of dose titration in the Open-label period
Arm/Group | MCI-196 (Double-blind Period) | Placebo (Double-blind Period)
Number analyzed (Participants) | 85 | 83
mg / dL | -0.04 (1.49) [-1.45 to -0.57] | 0.71 (1.71)

2. Secondary Outcome: Change From Baseline in Serum Phosphorus
Time Frame: 12 weeks (Week 0 to Week 12)
Population: ITT1 (The ITT1 population included all enrolled subjects who have taken at least one dose of study medication and have at least one central phosphorus value after the start of study medication.)
Measure: Mean (95% Confidence Interval); unit: mg/dL
Groups:
- MCI-196 (Open-label Period): 3, 6, 9, 12, or 15g/day as titrated (Week 0 -12)
Arm/Group | MCI-196 (Open-label Period)
Number analyzed (Participants) | 241
mg/dL | -1.54 [-1.80 to -1.28]

3. Secondary Outcome: Change From Baseline in PTH
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in Calcium
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Calcium x Phosphorus Ion Product
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Change From Baseline in Total Cholesterol
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Change From Baseline in LDL Cholesterol
Time Frame: 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Change From Baseline in HDL Cholesterol
Time Frame: 12 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Change From Baseline in VLDL Cholesterol
Time Frame: 12 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Change From Baseline in Triglyceride
Time Frame: 12 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Incidence of Adverse Events
Time Frame: 12 weeks (Week 0-12) and 4 weeks (Week 12-16)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks (Week 0-12) and 4 weeks (Week 12 - 16)
Description: Open-label Period is 12 weeks from Week 0 to Week 12. Double-Blind Period is 4 weeks after randomization at Week 12.
Groups:
- MCI-196 (Open-label Period): 3, 6, 9, 12, or 15 g/ day as titrated (Week 0-12)
- MCI-196 (Double-blind Period); Placebo (Double-blind Period): dose level at the end of dose titration in the Open-label period (Week 12-16)
  One subject who was randomized to placebo and another subject who was randomized to MCI-196 took both placebo and MCI-196 during the double-blind period. They have therefore been included in the MCI-196 group for the safety evaluation for the double-blind period.
Arm/Group | MCI-196 (Open-label Period) | MCI-196 (Double-blind Period) | Placebo (Double-blind Period)
Serious Adverse Events (participants affected / at risk) | 37/245 | 10/86 | 7/83
Other Adverse Events (participants affected / at risk) | 161/245 | 34/86 | 25/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MCI-196 (Open-label Period) (N=245) | MCI-196 (Double-blind Period) (N=86) | Placebo (Double-blind Period) (N=83)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 3 | 0 | 0
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Arteriovenous graft site infection (Infections and infestations) | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 2 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 1 | 0
Hypotension (Vascular disorders) | 3 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 2 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Colonoscopy abnormal (Investigations) | 1 | 0 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 3 | 0 | 0
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0
Superior vena caval occlusion (Vascular disorders) | 0 | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-196 (Open-label Period) (N=245) | MCI-196 (Double-blind Period) (N=86) | Placebo (Double-blind Period) (N=83)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 11 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3 | 1 | 1
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 6 | 0 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 2 | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 2 | 0 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 5 | 1 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 6 | 0 | 3
Influenza (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 2
Tooth infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 9 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0
Lymphangitis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Arteriovenous fistula site infection (Infections and infestations) | 2 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Eyelid infection (Infections and infestations) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 21 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 22 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 12 | 0 | 0
Vomiting (Gastrointestinal disorders) | 18 | 3 | 0
Abdominal discomfort (Gastrointestinal disorders) | 4 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 5 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 15 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 3 | 1 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Conduction disorder (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Chills (General disorders) | 3 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 6 | 3 | 1
Chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 6 | 1 | 0
Asthenia (General disorders) | 7 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 4 | 2 | 1
Influenza like illness (General disorders) | 1 | 0 | 0
Tenderness (General disorders) | 1 | 0 | 0
Face oedema (General disorders) | 3 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 4 | 1 | 0
Hypertension (Vascular disorders) | 6 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 10 | 1 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 3 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 4 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 2 | 0 | 0
Blood triglycerides increased (Investigations) | 2 | 0 | 0
Carbon dioxide decreased (Investigations) | 2 | 0 | 1
High density lipoprotein decreased (Investigations) | 2 | 0 | 0
Urine output decreased (Investigations) | 1 | 0 | 0
Very low density lipoprotein increased (Investigations) | 2 | 0 | 0
Vitamin D decreased (Investigations) | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood calcium decreased (Investigations) | 1 | 0 | 0
Blood parathyroid hormone increased (Investigations) | 2 | 0 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Calcium deficiency (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 0 | 1
Insomnia (Psychiatric disorders) | 5 | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Lip pain (Gastrointestinal disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Keloid scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1
Arteriovenous graft site infection (Infections and infestations) | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1 | 0
Bundle branch block (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 0 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1
Osteocalcin increased (Investigations) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other